CLINICAL TRIAL: NCT06574334
Title: Effect of Proprioceptive Exercises on Joint Pain and Quality of Life Among Geriatric Patients With Knee Osteoarthritis
Brief Title: Proprioceptive Exercises on Joint Pain and QoL Among Geriatric Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Hamdi Mahmoud, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KOA Geriatric
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: -Quasi experimental research design was used in this study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group received proprioceptive exercises (Experimental): - The study group included education about definition, components and benefits of proprioceptive exercises for geriatric patients with knee osteoarthritis in the first week. Also, was including proprioceptive exercises that included; One-leg balance, Toe walking, Heel walking, Cross-body leg swings, Blind advanced one leg balance and instructed them to do these 5 exercises (15-20 repetitions of each) per session, 5 day a week.
  Interventions: Procedure: Proprioceptive exercise
- the control group received routine exercise (Isometric exercise). (Experimental): the control group included education about definition, benefits and steps of isometric exercise that included participants taking the long sitting position. A role of towel was placed below the affected knee. The participants were then asked to press the towel down and hold it to one minute and then relax. This was repeated again for the other knee and (10-15 repetitions) per session, 5 day a week.
  Interventions: Procedure: Proprioceptive exercise

INTERVENTIONS:
Procedure: Proprioceptive exercise — * The first session was included an orientation to the exercises and its purpose to geriatric participants in the first week. Also, pretest was done in the first session before implementing exercises to assess geriatric KOA pain and QOL, each session started by revision about what was given during the previous session and the objectives of the next session.
  * The 2nd session about exercises.
  * The 3rd session for repetition of exercises to ensure that the patient has learned it well in the second week.
  * The 4th session after six weeks later (from wk. (3) to wk. (8) to make posttest after implementation session.
  * The 5th session after two-month later (from wk. (9) to wk. (16) to do follow up test.

SUMMARY:
Knee osteoarthritis, the disease of knee joint pain caused by joint degeneration, it is the commonest joint disease and had a negative effect on geriatric patients' quality of life (QoL). Proprioceptive exercise and isometric exercise have been recommended as suitable for reducing joint pain and improvement of quality of life in the geriatric patients.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA), known as degenerative joint disease of the knee. It is most common in the geriatric and is typically the result of wear and tear and progressive loss of articular cartilage. It happens when cartilage in knee joint breaks down. When this happens, the bones in knee joint rub together, causing friction that makes knees hurt, become stiff or swell. Knee OA is a painful condition and causes exhaustion in affected patients. Patients with this illness often complain of pain, decreased muscle strength, and joint instability. In addition, increased pain in knee OA patients also progressively worsen their quality-of-life. Proprioceptive activity in patients with knee OA gets limited or reduced and leads to reduced activities of daily living (ADLs). Joint proprioception is the ability of an individual to sense the joint position and movement. It encompasses the joint motion and joint position so proprioceptive exercises are being used for the strengthening of muscles around the knee joint. Thus, proprioceptive exercises are recommended exercise which significantly improved pain in knee OA patients which as results lead to improve quality of life. Quadriceps strengthening has been an important component of exercise program of knee osteoarthritis. This is because quadriceps weakness is the most presented finding among people with knee osteoarthritis. An isometric exercise is a form of exercise involving the static contraction of a muscle without any visible movement in the angle of the joint which lead to reduce joint pain and improving QoL in geriatric patients with knee osteoarthritis. The study sample (70) geriatric patients received proprioceptive exercises only, while the control group (70) geriatric patients received routine exercise (Isometric exercise) only.

ELIGIBILITY:
Inclusion criteria:

* Geriatric patients aged 60 years and above diagnosed with knee OA.
* Male and female geriatric patients.
* Alert and able to communicate.
* Mild and moderate knee OA (based on X-rays)

Exclusion criteria:

* Patients with advanced knee OA.
* Patients with end stage organ failure.
* Patients with cognitive impairment who will not be able to take active part in the study.
* Patients with neurological impairment or physical disability that interfere with their participation in the study.
* Patients with uncontrolled medical conditions.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of proprioceptive exercises on joint pain among geriatric patients with knee osteoarthritis | 3 months
  By using Visual Analog Scales (VAS):
Evaluate the effect of proprioceptive exercises on quality of life among geriatric patients with knee osteoarthritis | 3months
  By using 36 - Item Short-Form Health Survey (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt